CLINICAL TRIAL: NCT05093361
Title: Randomized Controlled Trial of Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5203108
Record Dates: First submitted 2018-12-10; First posted 2021-10-26 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-04

CONDITIONS: Hip Arthritis; Total Hip Arthroplasty (THA)
Keywords: Hip Arthritis; Total Hip Arthroplasty; THA; Conservative Treatment
MeSH Terms: interventions — Arthroplasty, Replacement, Hip; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative Treatment (Active Comparator): Total Hip Arthroplasty
  Interventions: Procedure: Total Hip Arthroplasty
- Conservative Treatment (Active Comparator): Physical therapy
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — Total Hip Arthroplasty for the treatment of hip arthritis.
  Arms: Operative Treatment
Procedure: Physical Therapy — Self-driven training according to the training plan instructed by physical therapist.
  Arms: Conservative Treatment

SUMMARY:
The purpose of this study is to compare the effect of total hip arthroplasty and conservative treatment to hip pain, to activities of daily life and to the quality of life in patients with hip osteoarthritis.

DETAILED DESCRIPTION:
The purpose of this randomized controlled study is to compare the effect of total hip arthroplasty and conservative treatment (that consists of self-driven exercises that physical therapists teach to the patients) to hip pain, to activities of daily life and to the quality of life in patients with hip osteoarthritis. Also the ill effects and cost effectiveness of total hip arthroplasty and conservative treatment are evaluated. Further more the aim is to investigate if total hip arthroplasty alleviates osteoarthritic pain in 12-month follow-up and if it enhances performance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Hip osteoarthritis that is in X-ray pictures ≥2 in Kellgren - Lawrence classification
* Primary osteoarthritis
* Patients symptoms of hip osteoarthritis are so severe, that an experienced orthopedist would suggest total hip arthroplasty as a treatment

Exclusion Criteria:

* Patients symptoms are so severe that total hip arthroplasty should be done within the next three months
* ASA > 3 (ASA physical status classification system)
* Normal contraindications to surgery
* Previous surgery to the same hip that has the osteoarthritis (including total hip arthroplasty, surgery for fracture, osteotomy, arthroscopy)
* The referring orthopedist has placed the patient in line for hip arthroplasty
* Secondary osteoarhritis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | From baseline to one year
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints.
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Physical functioning questions cover everyday activities such as stair use, standing up from a sitting or lying position, standing, bending, walking, getting in and out of a car, shopping, putting on or taking off socks, lying in bed, getting in or out of a bath, sitting, and heavy and light household duties. Higher scores indicate worse pain, stiffness, and functional limitations.
Harris Hip Score (HHS) | From baseline to one year
  The Harris Hip Score (HHS) is a clinician-based outcome measure frequently used for the evaluation of patients following a total hip arthroplasty.
  Four subscales make up HHS. The first is pain, which measures pain severity (44 points); function, which is made up of daily activities and gait (47 points); the absence of deformity, which is a subscale that measures hip flexion, adduction, internal rotation, leg length discrepancy and range of motion measures.(4 points), and range of motion (5 points).
  The survey has 10 question items and scores range from 0-100 with higher scores representing less dysfunction and better outcomes.

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Sub Score Pain | From baseline to one year
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints.
  The WOMAC measures five items for pain (score range 0-20). Higher scores indicate worse pain.
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Sub Score Stiffness | From baseline to one year
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints.
  The WOMAC measures two items for stiffness (score range 0-8). Higher scores indicate worse stiffness.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Sub Score Physical Function | From baseline to one year
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints.
  The WOMAC measures 17 items for functional limitation (score range 0-68). Physical functioning questions cover everyday activities such as stair use, standing up from a sitting or lying position, standing, bending, walking, getting in and out of a car, shopping, putting on or taking off socks, lying in bed, getting in or out of a bath, sitting, and heavy and light household duties. Higher scores indicate worse functional limitations.
30s Chair Stand Test | From baseline to one year
  How many times a patient can stand up and sit down on a chair in 30 seconds. Higher scores mean a better outcome.
40m Fast-paced Walk Test | From baseline to one year
  How fast can a patient walk 40 meters measured in seconds. Lower scores mean a better outcome.
Stair Climb Test | Baseline to one year
  The time (in seconds) it takes to ascend and descend a flight of stairs. Lower scores mean a better outcome.
Grip Strength | Baseline to one year
  Maximum grip strength with dominant hand. Three squeezes are measured with Jamar Hand Dynamometer. Higher scores mean a better outcome. Force is measured in kilograms.
Short Form 36 Health Survey Questionnaire (SF-36) | Baseline to one year
  The 36-Item Short Form Survey (SF-36) is an self-reported measure of health. It stems from a study called the Medical Outcomes Study.
  It comprises 36 questions which cover eight domains of health:
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions
  Patients or individuals are asked to fill out the questionnaire (tick boxes) by themselves and then it is scored by a clinician or researcher.
  Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to high QOL.
painDetect | Baseline to one year
  painDETECT is a nine-item questionnaire that consists of seven sensory symptom items for pain that are graded from 0= never to 5= strongly, one temporal item on pain-course pattern graded -1 to +1, and one spatial item on pain radiation graded 0 for no radiation or +2 for radiating pain. A total score that ranges from -1 to 38 can be calculated from the nine items, with higher scores indicating higher levels of neuropathic pain.
BMI | Baseline to one year
  Body Mass Index (BMI). Weight and height will be combined to report BMI in kg/m^2.
Use of pain medication | Baseline to one year
  Rate of pain medication use (paracetamol, NSAID and opioid pain medication) in four stage rating.
  1. Not at all
  2. Few days a month
  3. Few days a week
  4. Daily
Training diary | Baseline to one year
  Patients keep a record of the training they do at home. The exercises are taught by the physical therapists and patients mark the number of days per week, that they have done the exercises.
Range of motion in hip extension | Baseline to one year
  Measurement of hip extension in side lying position. Measurement is done by physical therapist with a goniometer and it is reported in degrees.
Range of motion in hip flexion | Baseline to one year
  Measurement of hip flexion in side lying position. Measurement is done by physical therapist with a goniometer and it is reported in degrees.
Range of motion in hip inner rotation | Baseline to one year
  Measurement of hip inner rotation in supine position. Measurement is done by physical therapist with a goniometer and it is reported in degrees.
Range of motion in hip outer rotation | Baseline to one year
  Measurement of hip inner rotation in supine position. Measurement is done by physical therapist with a goniometer and it is reported in degrees.
Leg length discrepancy | Baseline to one year
  Leg length is measured from the highest point of ileum. Measurement is done by physical therapist and reported in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Aapo Talonpoika, Principal Investigator — Kuopio University Hospital; Jari Arokoski, Study Director — Kuopio University Hospital and Helsinki University Hospital; Lauri Karttunen, Principal Investigator — Kuopio University Hospital; Hannu Luomajoki, Study Director — Zürcher Hochschule für Angewandte Wissenschaften ZHAW Departement Gesundheit, Institut für Physiotherapie; Jukka Huopio, Study Director — Kuopio University Hospital; Antti Jaroma, Study Director — Kuopio University Hospital; Joonas Sirola, Study Director — Kuopio University Hospital; Heikki Kröger, Study Chair — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland